CLINICAL TRIAL: NCT05211648
Title: COOL-BP Study: Continuous Versus Occasional Blood Pressure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OBPM_Remote2021
Record Dates: First submitted 2021-12-23; First posted 2022-01-27 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This is a prospective open-label single arm study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Patients with Aktiia bracelet (Experimental): This is a prospective open-label single arm study. Study participants will wear the Aktiia bracelet for 6 months and will continue in parallel the procedures of the Remote Hypertension Program.
  Interventions: Device: Aktiia Bracelet

INTERVENTIONS:
Device: Aktiia Bracelet — Aktiia Bracelet is a CE-marked medical device that will be used in accordance with its instructions for use. The optical signals at the wrist are recorded non-invasively by means by the Aktiia bracelet. The Blood Pressure measurements are further determined from these optical signals and are compared to weekly and monthly Blood Pressure averages measured manually by traditional Home Blood Pressure Monitoring.

SUMMARY:
The COOL-BP study is part of the Remote Hypertension Program and will investigate the data provided by Aktiia Bracelet (a cuffless Blood Pressure monitor at the wrist) when integrated into the Remote Hypertension Program.

The COOL BP study aims to compare weekly and monthly Blood Pressure averages measured manually by traditional Home Blood Pressure Monitoring to those measured automatically by the Aktiia bracelet.

DETAILED DESCRIPTION:
This is a prospective open-label single arm study. The investigational device of this study is the Aktiia Bracelet device. Aktiia Bracelet is a non-invasive blood pressure (BP) monitor intended to track systolic and diastolic Blood Pressure trends. The Aktiia Bracelet can also measure heart rate.

Participants who consent to participate in COOL-BP will be shipped an Aktiia device to participants' residence.

For 6 months, patient will continue the procedures of the Remote Hypertension Program in parallel to wearing the Aktiia Bracelet. The Remote Hypertension Program is run remotely according to a clinical algorithm, where study navigators contact patients at regular intervals and monitor symptoms by regular phone calls; laboratory tests are obtained to ensure safety of the protocol's prescribed medications. Any symptoms will be evaluated by the program nurse practitioner or physician and managed per standard of care. During the study, the patient completes several surveys to give opinion on Aktiia product versus Home Blood Pressure Monitoring.

Following six months of using the Aktiia.product, the participant's participation in this study will end. Participants continued participation in the Remote Hypertension Program will depend on whether participants have met the blood pressure goals outlined in that program.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in written and spoken English
* Already enrolled in the Remote Hypertension Program
* Average of last 3 office blood pressures >140/90 mm Hg in last 18 months OR Last office blood pressure >140/90 mm Hg in last 6 months OR Referred by MD and last 1 blood pressure >130/80 mm Hg
* Own an iPhone

Exclusion Criteria:

* Tachycardia (heart rate at rest > 120bpm)
* Atrial fibrillation, persistent
* Severe heart failure (LVEF<35%)
* Pheochromocytoma
* Raynaud's disease
* Trembling and shivering
* Known pregnancy
* Breastfeeding
* Arteriovenous fistula
* Arm amputation
* Exfoliative skin disease
* Lymphoedema
* Known allergy to silicone
* Not Massachusetts resident
* Last MGB office visit >3 years
* No-MGB provider
* Terminal medical condition
* CKD 4-5 (eGFR ≤ 30 mL/mn)

Ages: 26 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Diastolic and Systolic Pressures differences between weekly Diastolic and Systolic pressures averages provided by Home Blood Pressure Monitoring and by Aktiia 24h data. | 6 months
  Diastolic and Systolic Pressures are measured weekly manually by traditional Home Blood Pressure Monitoring and continuously with the Aktiia bracelet.
Diastolic and Systolic Pressures differences between monthly Diastolic and Systolic pressures averages provided by Home Blood Pressure Monitoring and by Aktiia 24h data. | 6 months
  Diastolic and Systolic Pressures are measured monthly manually by traditional Home Blood Pressure Monitoring and continuously with the Aktiia bracelet.

SECONDARY OUTCOMES:
Diastolic and Systolic Pressures Circadian profiles | 6 months
  Analysis of the evolution of Diastolic and Systolic Pressures circadian profiles of each patient during the study.
Quality of life surveys | 6 months
  Participants complete the same survey at Day 30, Day 60 and Day 180 to give a feedback on participants' satisfaction and comfort regarding Aktiia product compared to Home Blood Pressure monitoring. Part of answers to surveys are based on satisfaction scales from 0 to 10 where 0 = "bad" and 10 = "good".

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fisher, MD, Principal Investigator — Harvard Medical School Boston MA
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No